CLINICAL TRIAL: NCT01693549
Title: Phase II Study of Cabazitaxel as 2nd Line Treatment in Patients With HER-2 Negative Metastatic Breast Cancer Previously Treated With Taxanes
Brief Title: Study of Cabazitaxel in Patients With Metastatic Breast Cancer Previously Treated With Taxanes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE 11B/11; 2011-003625-97 (EudraCT Number)
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: HER-2 negative; Metastatic breast adenocarcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — cabazitaxel; XRP6258

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel (Experimental): Cabazitaxel(XRP6258) will be administered on day 1 of each cycle, every 21 days, at a dose of 25 mg/m² by i.v. route in 1 hour. Treatment can be continued until patient's consent withdrawal, intolerable toxicity or documented disease progression.
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel
  Other Names: Jevtana; XRP6258

SUMMARY:
The purpose of this study is to determine whether cabazitaxel is effective in the treatment of metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female patients aged 18 to 75 years
* Patients must have received 1st-line chemotherapy for locally recurrent / metastatic disease
* Prior taxane-containing treatment (paclitaxel, docetaxel or nab-paclitaxel), either for advanced disease or as neoadjuvant/adjuvant chemotherapy. In case of early relapse (relapse during neoadjuvant/adjuvant chemotherapy or disease-free interval less than 6 months), neoadjuvant/adjuvant chemotherapy will be considered as 1st-line treatment
* Diagnosis of HER-2 negative (HER-2 <2+ by immunohistochemistry and/or FISH or CISH negative) metastatic breast adenocarcinoma confirmed by the pathology department of the enrolling institution
* Eastern Cooperative Oncology Group performance status (PS) of 0-1
* Life expectancy of at least 12 weeks
* Measurable disease by the Response Criteria in Solid Tumors 1.1 (RECIST 1.1) method (at least one measurable lesion)
* Laboratory values within the specified ranges within 1 week of study enrolment:

  1. Hemoglobin ≥ 9.0 g/dL
  2. Absolute neutrophil count of ≥ 1.5 x 10^9/L
  3. Thrombocyte count of ≥ 100 x 10^9/L
  4. Serum creatinine ≤ 1.5 upper limit of normal (ULN). If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance <60 mL/min should be excluded
  5. SGOT (AST), SGPT (ALT) ≤ 2.5 x ULN and alkaline phosphatase ≤ 2.5 x ULN, total bilirubin ≤ ULN (the same limits also refer to patients with liver metastases)
* Previous treatment for loco-regional disease is allowed, including surgical procedures or palliative radiotherapy (such treatments must have been completed at least 4 weeks before enrolment)
* Compliance of the patient regarding scheduled visits, treatment plan, laboratory tests and other procedures of the study.
* The enrolment of patients with controlled brain metastases is allowed (metastases that have been treated with radiotherapy and remained stable for at least 4 weeks following the completion of radiation treatment)

Exclusion Criteria:

* Patients that have received more than one lines of chemotherapy for locally recurrent/metastatic disease
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a wash-out period of two weeks is necessary for patients who are already on these treatments)
* Patients with CTC grade 2 or greater neuropathy at baseline
* Diagnosis of spinal cord compression or carcinomatous meningitis
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
* Patients with clinically significant cardiac disease (e.g. congestive heart failure, unstable angina, myocardial infarction) within 6 months from study entry
* Any other significant acute or chronic medical or psychiatric condition or abnormal laboratory finding which, according to the investigator's opinion, could result in excessive danger, regarding the participation of the patient in the study.
* Psychiatric disorders or other conditions rendering the subject incapable of complying with the requirements of the protocol
* Any concurrent active malignancy other than non-melanoma skin cancer or in situ carcinoma of the cervix
* Concurrent administration of other investigational treatments and/or anti-neoplastic agents
* Pregnancy or lactation. Patients should be surgically sterile or post-menopausal or they must agree to use adequate contraceptive methods during study period. For all patients of childbearing potential a serum or urine pregnancy test is needed. The definition of effective contraceptive methods will be based on the investigator's opinion.
* History of severe hypersensitivity reaction (≥grade 3) to docetaxel or polysorbate 80 containing drugs

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-09; Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR). | At an average of 24 months for each patient

SECONDARY OUTCOMES:
Duration of response. | From the time measurement criteria are first met for partial or complete response until the first date of documented progressive disease or death from any cause without prior documentation of progression assessed up to 30 months.
Evaluation of progression-free survival (PFS) | From study entry until the first date of documented progressive disease (PD) or death from any cause without prior documentation of progression, assessed up to 30 months.
Evaluation of overall survival (OS) | Defined as the time in months from study entry until the time of death, assessed up to 30 months.
Assessment of safety and tolerability. | Evaluation of Adverse Events will be performed every 21 days (per cycle) during treatment assessed up to 30 months.
  Distribution of adverse events according to severity grade.
Value of prognostic and/or predictive biomarkers measured in tissue and blood samples | Tumor blocks and blood DNA will be collected at study entry and plasma at study entry, on week 3 and week 6 of treatment.
  βΙ,βΙΙ,βΙΙΙ,βIVb, βV-tubulin isotypes,HIF1α,microtubule-associated proteins such as Tau,MAP2,MAP4 & microtubule-sequestering proteins such as stathmin, will be assessed. Moreover, evaluation of p53,BCL2,BIM,γ-actin,LIMK2, TGFBI,Aurora-A,as well as the expression of the enzyme CYP3A and multidrug transporters such as P-glycoprotein. The abovementioned factors will be assessed by immunohistochemistry at the protein level and by quantitative real-time PCR at the RNA level.
  Also, given the clinical significance of the anti-angiogenic effects of cytotoxic chemotherapy,we will investigate the effect of treatment on surrogate biomarkers of angiogenesis, such as VEGF-A as well as the effect of chemotherapy on kinetics of soluble biomarkers,using ELISA.
  In addition,genetic polymorphisms in drug-metabolizing enzymes and drug transporters, such as the CYP3A and ABCB1 genes, will be explored in blood DNA and their association with the toxicity and efficacy of cabazitaxel will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Angelos Koutras, MD, Study Chair — Division of Oncology,Dept of Internal Medicine,University Hospital of Patras
Locations (17):
- Greece (17):
  - Dept of Medical Oncology, 251 General Air Force Hospital, Athens
  - 2nd Dept of Medical Oncology, General Hospital of Athens "Hippokratio", Athens
  - Oncology section, Dept of Clinical Therapeutics, General Hospital of Athens "Alexandra", Athens
  - Division of Oncology, 2nd Dept of Internal Medicine, Propaedeutic, University Hospital "Attikon", Athens
  - 2nd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens
  - 3rd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens
  - 3rd Dept of Medical Oncology, Hygeia Hospital, Athens
  - 1st Dept of Medical Oncology, Metropolitan Hospital, Athens
  - 2nd Dept of Medical Oncology, Metropolitan Hospital, Athens
  - 2nd Dept of Medical Oncology, Agios Savvas Cancer Hospital, Athens
  - Oncology Dept., General Hospital of Chania "Agios Georgios", Chania
  - Dept of Medical Oncology, University Hospital of Heraklion, Heraklio
  - Dept of Medical Oncology, Ioannina University Hospital, Ioannina
  - General Hospital of Patra "Agios Andreas", Pátrai
  - Division of Oncology, Dept of Internal Medicine, University Hospital of Patras, Rio, Patras
  - Dept of Medical Oncology, Papageorgiou General Hospital, Thessaloniki
  - Dept of Medical Oncology, Thermi Clinic S.A, Thessaloniki